CLINICAL TRIAL: NCT07342426
Title: Comparison of the Effects of High and Low Dose High-intensity Laser Therapy in Patients With Lateral Epicondylitis
Brief Title: High and Low Dose High-intensity Laser Therapy Lateral Epicondylitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20250361
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lateral Epicondylitis; High Intensity Laser Therapy; Tennis Elbow; High Intensity Laser
Keywords: treatment
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Conrol group (Placebo Comparator): Placebo high intensity laser therapy with Infarred ray and Transcutaneous electrical nerve stimulator therapy
  Interventions: Device: Infarred ray therapy system; Device: Transcutaneous electrical nerve stimulator
- Low dosage group (Experimental): Low dosage High intensity laser with Infarred ray and Transcutaneous electrical nerve stimulator therapy
  Interventions: Device: High intensity laser therapy; Device: Infarred ray therapy system; Device: Transcutaneous electrical nerve stimulator
- High dosage group (Experimental): High dosage High intensity laser therapy with Infarred ray and Transcutaneous electrical nerve stimulator therapy
  Interventions: Device: High intensity laser therapy; Device: Infarred ray therapy system; Device: Transcutaneous electrical nerve stimulator

INTERVENTIONS:
Device: High intensity laser therapy — Using high-intensity laser therapy applying on the affected area.
  Arms: High dosage group; Low dosage group
Device: Infarred ray therapy system — Using infarred ray therapy applying on affected area for 15 minutes.
Device: Transcutaneous electrical nerve stimulator — Using transcutaneous electrical nerve stimulator on the affected area fior 15 minutes.

SUMMARY:
High-intensity laser therapy has gained increasing attention in recent years as a therapeutic modality. It is a non-invasive treatment that can reduce pain, increase local blood circulation, and promote tissue repair. The higher energy output of high-intensity laser therapy also have deeper tissue penetration. Several studies have investigated the effects of high-intensity laser therapy on lateral epicondylitis, and the existing literature indicates that, compared with other treatment modalities, high-intensity laser therapy is more effective in improving pain and quality of life in patients with lateral epicondylitis.

However, the dosage, duration, and treatment frequency applied in previous studies vary considerably. The therapeutic effects of high-intensity laser therapy may therefore be influenced by treatment dosage. Consequently, the purpose of this study is to compare the effects of two different dosages of high-intensity laser therapy on patients with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with lateral epicondylitis by physician
2. Disease duration of less than three months
3. Adults aged above 18 years with full decision-making capacity

Exclusion Criteria:

1. Patients who have received treatments other than standard treatment to the affected area within past three months
2. Patients with contraindication for rehabilitation therapy

   1. Photosensitivity
   2. Sensory impairment
   3. Implanted cardiac pacemaker
   4. Pregnancy
   5. Malignancy
3. Patients with a history of surgery on the affected elbow
4. Patients with cervical radiculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | From enrollment to the end of treatment at 4 weeks
  Using visual analog scale to measure pain intensity. Score from 0 to 10. Score 0 means no pain and score 10 indicates highest pain.

SECONDARY OUTCOMES:
Grip strength | From enrollment to the end of treatment at 4 weeks
  Using dynanometer to measure grip strength
Quality of life | From enrollment to the end of treatment at 4 weeks
  Using Quick disabilities of the Arm, Shoulder, and hand scale (also known as Quick DASH) to measure quality of life of participants. Scale contains 11 questions. Each question scored from 1 to 5, higher score indicates higher degree of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- TSAI CHENG-TAO Physical Therapy Clinic, Kaohsiung City, Taiwan